CLINICAL TRIAL: NCT04725994
Title: An Open-Label, International, Multicenter, Phase 1b/2a Study to Assess the Safety, Tolerability, and Efficacy of IDX-1197 in Combination with XELOX (Capecitabine and Oxaliplatin) or Irinotecan in Patients with Advanced Gastric Cancer
Brief Title: Study to Assess the Safety, Tolerability, and Efficacy of IDX-1197 in Combination with XELOX or Irinotecan in Patients with Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Idience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ID-VDP-103
Record Dates: First submitted 2021-01-13; First posted 2021-01-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer
Keywords: 1197; IDX-1197; venadaparib
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Other)
  Interventions: Drug: IDX-1197+XELOX
- Group 2 (Other)
  Interventions: Drug: IDX-1197+Irinotecan

INTERVENTIONS:
Drug: IDX-1197+XELOX — The dose levels will be escalated following a 3+3 dose escalation scheme.
  Arms: Group 1
Drug: IDX-1197+Irinotecan — The dose levels will be escalated following a 3+3 dose escalation scheme.
  Arms: Group 2

SUMMARY:
This is an open-label, Phase 1b/2a study to evaluate the safety and tolerability of IDX-1197 and determine the MTD and RP2D in combination with XELOX or irinotecan in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Group 1, patients with treatment-naïve recurrent or advanced metastatic gastric cancer including gastroesophageal junction or upper part of the stomach.
* Group 2, patients with recurrent or advanced metastatic gastric cancer including gastroesophageal junction or upper part of the stomach, who were treated ≥2 times with palliative chemotherapy before screening.
* At least 1 evaluable lesion for the dose escalation part and at least 1 measurable lesion according to RECIST v1.1 for the dose expansion part.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Group 2 Part C, patients should have UGT1A1 genotype tested during or prior to screening.

Exclusion Criteria:

* Symptomatic central nervous system or uncontrolled brain metastasis
* Carcinomatous meningitis or its history.
* For Group 1, patients who are HER 2 positive.
* Any other concurrent uncontrolled illness including, but not limited to, active or ongoing symptomatic infection requiring IV antibiotic treatment, uncontrolled diabetes, hepatic, renal, or respiratory illness.
* Severe or unstable angina, myocardial infarction or ischemia, symptomatic congestive heart failure, arterial or venous thromboembolism requiring coronary artery bypass graft or stent within the past 6 months or clinically significant cardiac dysrhythmia or New York Heart Association class II ~ IV heart disease within 6 months of randomization.
* Uncontrolled hypertension
* Immunocompromised patients, such as patients known to be serologically positive for HIV.
* Patients with known active Hepatitis B or C infection.
* Patients with known active or symptomatic pneumonitis, or history of non-infectious pneumonitis requiring steroids.
* Diagnosis of a myelodysplastic syndrome/acute myeloid leukemia or its suspicious characteristics.
* Any unresolved clinically significant Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 toxicity
* Resting ECG with measurable QTcF > 470 msec on 2 or more time points within a 24-hour period or family history of long QT syndrome.
* Current use of a cytochrome P3A4 inhibitor or inducer and strong uridine diphosphate (UDP)-glucuronosyltransferase 1A1 (UGT1A1) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) | through study completion (Up to 12 months)
  To determine the MTD and RP2D of IDX-1197 when given in combination with XELOX or Irinotecan. This will be accomplished by the standard 3+3 dose escalation design. If 2 of the 3 to 6 patients in a particular dose level experience a DLT, the dose escalation should be stopped at this dose level, and the MTD will be determined.
Dose Limiting Toxicities (DLTs) | during the first 21-day cycle for Group 1 and through first 2 cycles (14 days each) for Group 2
  Occurrence of DLTs

CONTACTS AND LOCATIONS:
Locations (14):
- United States (4):
  - USC Norris Comp. Cancer Ctr Hospital, Los Angeles, California
  - Hematology Oncology Clinic Baton Rouge / Sarah Cannon, Baton Rouge, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Astera Cancer Care, East Brunswick, New Jersey
- China (3):
  - Beijing Cancer Hospital, Beijing
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Shanghai East Hospital, Shanghai
- South Korea (7):
  - Dong-A University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided